CLINICAL TRIAL: NCT04705129
Title: A Phase II Study on the Safety and Efficacy of Zanubrutinib Combined With Tislelizumab in the Treatment of Relapsed/Refractory Primary Mediastinal Large B-cell Lymphoma and Epstein-Barr Virus-positive Diffuse Large B-cell Lymphoma
Brief Title: Zanubrutinib Combined With Tislelizumab in the Treatment of r/r PMBCL and EBV+ DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-PMBCL-1
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Primary Mediastinal Large B Cell Lymphoma; EBV-Positive DLBCL, Nos
Keywords: Primary Mediastinal Large B Cell Lymphoma; EBV-Positive DLBCL, nos; targeted therapy
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — zanubrutinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zanubrutinib+Tislelizumab (Experimental): Zanubrutinib 160mg Bid, D1-21, po；Tislelizumab 200mg, D1, ivgtt
  Interventions: Drug: Zanubrutinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Zanubrutinib — 160mg Bid, D1-21, po
Drug: Tislelizumab — 200mg, D1, ivgtt

SUMMARY:
The study is to investigate the safety and efficacy of Zanubrutinib combined with Tislelizumab in the treatment of relapsed/refractory primary mediastinal large B-cell lymphoma and Epstein-Barr Virus-positive diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
R-CHOP regimen is the first-line therapy in DLBCL which greatly improved the efficacy of diffuse large B-cell lymphoma (DLBCL) and achieved good long-term survival. However, among DLBCL patients treated with R-CHOP, EBV+ had a lower 5-year OS than EBV- patients (65% vs 82%). For primary mediastinal large B-cell lymphoma (PMBCL), although the initial treatment has a better prognosis than DLBCL, there are still 10% to 30% of PMBCL patients with primary refractory or relapsed disease, and the prognosis is poor.

Zanubrutinib combined with Tislelizumab has been proved efficient in relapsed or refractory NHLs, with ORR rate 37%, CR rate of 16.7%. This phase II, prospective, open-label, single-arm study will evaluate the efficacy and safety of Zanubrutinib combined with Tislelizumab in the treatment of relapsed/refractory primary mediastinal large B-cell lymphoma and Epstein-Barr Virus-positive diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diffuse large B-cell lymphoma, EBV positive and primary mediastinal large B-cell lymphoma
* Have received at least one prior standard therapy line including Rituximab and anthracyclines.
* Age≥18
* ECOG 0,1,2
* Imaging accessible lesions
* Life expectancy>3 months
* Informed consented

Exclusion Criteria:

* Have received systemic or local treatment including chemotherapy within three weeks before enrollment
* Chronic or active infectious diseases that require systemic antibiotics, antifungals or antiviral therapy
* Lab at enrollment (Unless caused by lymphoma) : Neutrophile<1.0*10^9/L , Hemoglobin<80g/L, Platelet<50*10^9/L, ALT or AST >2*ULN,AKP or bilirubin >1.5*ULN Creatinine>1.5*ULN
* Other uncontrollable medical condition that may that may interfere the participation of the study Not able to comply to the protocol for mental or other unknown reasons
* HIV infection
* If HbsAg positive, should check HBV DNA, DNA positive patients cannot be enrolled. If HBsAg negative but HBcAb positive (whatever HBsAb status), should check HBV DNA, DNA positive patients cannot be enrolled
* Previously received BTK inhibitor or anti-PD-1/PD-L1 treatment
* History of active autoimmune disease or severe autoimmune disease
* Need to be given corticosteroids (dose equivalent to prednisone >20 mg/day) or other immunosuppressive agents within 14 days before the study drug administration
* A history of interstitial lung disease or non-infectious pneumonia, except for those caused by radiotherapy
* Need strong cytochrome P450 (CYP) 3A inhibitor or inducer drug treatment
* Received live vaccination within 28 days before the first dose of study drug
* Patients who can receive hematopoietic stem cell transplantation, and if the subject has received allogeneic stem cell transplantation within 6 months before the first administration of the study drug or has active graft-versus-host disease requiring continuous immunosuppressive therapy
* Have received any experimental drug within 28 days, or the toxicity of any previous chemotherapy has not been relieved to ≤ Grade 1
* History of malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, unless recovered for at least 2 years
* Have a history of other active malignancies within 2 years before entering the study, excluding cervical cancer in situ, local basal cell or squamous cell skin cancer that has been cured by adequate treatment; or the previous malignant tumor is localized and has undergone local radical treatment Treatment (surgery or other forms)
* Pregnant or nursing period
* Men or women who are fertile but refuse to take appropriate contraceptive measures, unless they have been surgically sterilized

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 21 days after 6 cycles of treatment (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
progression free survival | 2 year
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
overall survival | 2 year
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event. of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Up to 30 days after completion of study treatment
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events

OTHER OUTCOMES:
The significance of biomarkers in tissue and plasma including cfDNA, PD-1,PD-L1 | through study completion，an average of 2 years
  Dynamic change of the expression of PD-1, PD-L1

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, PhD, MD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No